CLINICAL TRIAL: NCT07007975
Title: The Effect of Web-based Gynecological Cancer Awareness on Married Women's Gynecological Cancer Awareness and Healthy Lifestyle Behaviors
Brief Title: The Effect of Web-based Education on Gynecological Cancer Awareness and Healthy Life Behaviors
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, DERYA YÜKSELEN EROL, PhD Student, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DYUKSELENEROL
Record Dates: First submitted 2025-05-25; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy Women

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web based training (Experimental): Web-based training will be given to experimental group and the results of the training will be evaluated
  Interventions: Behavioral: Web based training
- control group (No Intervention): Participants in this group will not be provided with training

INTERVENTIONS:
Behavioral: Web based training — This group will receive information about healthy lifestyle behaviors and gynecological cancer awareness.
  Arms: Web based training

SUMMARY:
There are cross-sectional or quasi-experimental studies in the literature on gynecological cancer awareness, but there are no fully experimental studies. The study we will conduct will use a control group and will be a fully experimental study. Thus, it is thought to contribute more to the field. The purpose of the study is to determine the effect of gynecological cancer education given to married women on their gynecological cancer awareness and healthy living behaviors.

DETAILED DESCRIPTION:
The aim of the study was to determine the effect of web-based gynecological cancer education on gynecological cancer awareness and healthy life behaviors of married women. For this purpose, participants were divided into two groups and web-based education was given to the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20-65
* Being open to communication
* Being literate
* Being able to use the internet
* Having a smart phone or computer

Exclusion Criteria:

* Being pregnant
* Being breastfeeding
* Not being able to use a website
* Not having watched all the videos on the website
* Having a history of gynecological cancer in oneself or in one's family

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women participated
Enrollment: 120 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
Gynecological cancer awareness scale | 4 weeks
  Preliminary test results received. The minimum score that can be obtained from the scale is 41, the maximum score is 205. The pre-training scale score average of the experimental group is 90.97.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagül Y Yağmur, Study Director — Inonu University
Locations (1):
- Family Health Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Scale results will be shared.
Supporting Information: SAP
Time Frame: It will be accessible in March 2025. It will be accessible for 6 months.
Access Criteria: Those working in the field of nursing will be able to access it.